CLINICAL TRIAL: NCT03716856
Title: Clinical Study of Redirected Autologous T Cells With a BCMA-targeted Chimeric Antigen Receptor in Patients With Refractory or Relapsed Multiple Myeloma
Brief Title: Clinical Study of CAR-BCMA T in Patients With Refractory or Relapsed Multiple Myeloma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: CARsgen Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CG6003
Record Dates: First submitted 2018-09-27; First posted 2018-10-23 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Refractory or Relapsed Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-BCMA T cells (Experimental): In this study, autologous T cells transduced with a BCMA-targeted chimeric antigen receptor (CAR-BCMA T cells) are used to treat patients with refractory or relapsed multiple myeloma.
  Route of administration: Intravenous injection.
  Lymphodepletion conditioning:
  Lymphodepletion will be conducted several days prior to CAR-BCMA T cells infusion.
  A combination of fludarabine and cyclophosphamide will be used for lymphodepletion.
  Interventions: Genetic: CAR-BCMA T cells; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Genetic: CAR-BCMA T cells — Single dose of CAR-BCMA T cells will be infused, and classic "3+3" dose escalation will be applied.
  Other Names: BCMA-redirected autologous T cells
Drug: Fludarabine — Fludarabine is used for lymphodepletion.
Drug: Cyclophosphamide — Cyclophosphamide is used for lymphodepletion

SUMMARY:
A single arm, open-label pilot study is designed to determine the safety, efficacy and cytokinetics of CAR-BCMA T cells in patients with BCMA-positive refractory or relapsed multiple myeloma.

DETAILED DESCRIPTION:
This study is designed to determine the safety, tolerability and engraftment potential of anti-BCMA lentivirus-transduced autologous T cells in patients with refractory or relapsed multiple myeloma.

Primary objectives:

1. Determine the safety and tolerability of CAR-BCMA T cells (autologous T cells transduced with chimeric antigen receptors recognizing BCMA) in patients with refractory or relapsed multiple myeloma.
2. Observe the cytokinetics of CAR-BCMA T cells.

Secondary objectives:

1. Observe the anti-tumor response of CAR-BCMA T cells to refractory or relapsed multiple myeloma (evaluated by diagnostic criteria International Myeloma Working Group (IMWG2014 version) as CR, sCR, ICR, MCR or VGPR).
2. Make an evaluation on the distribution and in vivo survival of CAR-BCMA T cells in peripheral blood, lymph node, and bone marrow.
3. Observe the immunogenicity of CAR-BCMA T cells, and determine if there is anti-BCMA scFv cellular immune response and anti-BCMA scFv humoral immune response.
4. Observe the change of T cell subsets relative to CAR-BCMA T。 (Tcm, central memory T lymphocytes; Tem, effector memory T lymphocytes; Treg, regulatory T lymphocytes).

ELIGIBILITY:
Inclusion Criteria：

* Patients aged between 18 ~ 70 with relapsed or refractory multiple myeloma.
* Bone marrow sample is confirmed as BCMA-positive by flow cytometry or pathological examination.
* Patients with relapsed or refractory multiple myeloma who meet the following conditions:

  1. Curative efficacy is little or disease progressed after 2 courses of standard treatment regimen;
  2. Disease relapsed after chemotherapy or HSCT. Curative efficacy is little or disease progressed after 2 courses of original treatment regimen;
  3. More than 60 days between last treatment and disease progression;
  4. Autologous or allogeneic SCT is not available at present, or patient refuses to receive SCT;
  5. No response to treatment is defined according to International Myeloma Working Group 2014 version as not achieving CR (including CR, sCR, ICR, MCR) or PR (including VGPR, PR, MR) after 2 consecutive cycles of treatment with current therapy, and the interval between the 2 cycles is no more than 60 days. Disease progression is defined as per 《Chinese Guidelines for Diagnosis and Treatment of Multiple Myeloma》 (Revision in 2015). At least one of the following conditions should be met:Serum M-protein increases ≥ 25% (absolute increase should be ≥ 5 g/L); If serum M protein is ≥ 50 g/L at baseline, increase of serum M protein can be ≥ 10 g/L; Urine M-protein increases ≥ 25% (absolute increase should be ≥ 200 mg/24 h); If the serum and urine M-protein are not detectable, a ≥ 25% increase in the difference between involved and uninvolved FLC levels is required (absolute increase should be ≥ 100 mg/L); Bone marrow plasma cell percentage increases ≥ 25% (absolute increase should be ≥ 10%); Size of existing bone lesions or soft tissue plasmacytomas increases by ≥ 25%, or development of new lytic bone lesions or soft tissue plasmacytomas; Development of hypercalcemia that can be attributed to plasma cell proliferative disorder (corrected calcium is > 2.8 mmol/L or 11.5 mg/dL); Disease progression must be confirmed by 2 sequential assessments.
* Expected survival > 12 weeks.
* Disease is measurable, and at least one of the following conditions should be satisfied:
* Serum M-protein is ≥ 10 g/L;
* 24-hour urine M-protein is ≥ 200 mg;
* Serum FLC is ≥ 5 mg/dL;
* Plasmacytomas that can be evaluated by tests or imaging;
* Bone marrow plasma cell percentage is ≥ 20%.
* ECOG scores 0 - 1.
* Adequate venous access for apheresis and venous blood sampling, and no other contraindications for leukapheresis.
* WBC ≥ 1.5×10^9/L;PLT ≥ 45×10^9/L; Hb≥9.0g/dL
* Serum creatinine ≤ 1.5 ULN.
* ALT ≤ 2.5 ULN;AST ≤ 2.5 ULN. The above lab results should not include those obtained from continuous supportive treatment that is ongoing.

Exclusion Criteria:

Patients with any of the following conditions are not eligible for this study.

* Pregnant or lactating women.
* HIV positive, or HCV positive
* Uncontrolled active infection, including active tuberculosis and HBV DNA copies ≥ 1×10^3 copies/mL.
* Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary.
* Allergic to immunotherapies and related drugs.
* Patients with heart disease for which treatment is needed or with poorly controlled hypertension.
* Hyponatremia: serum sodium level < 125 mmol/L.
* Baseline serum potassium < 3.5 mmol/L (taking potassium supplements before participating in the study to raise potassium level is acceptable).
* Previous treatment with chemoradiotherapy, local treatment ,immunotherapy and tumor-targeting drug conducted 2 weeks prior to participation in this study or blood collection.
* Patients have undertaken immunosuppressor for graft-versus-host disease (GVHD) within 4 weeks before participation in this study or blood collection, or the patient is diagnosed with acute or chronic GVHD.
* Other severe disease that may restrain patients from participating in this study (e.g. diabetes, severe cardiac dysfunction, myocardial infarction or unstable arrhythmias or unstable angina in recent 6 months, gastric ulcer, active autoimmune disease, etc.).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2020-06-23 (Actual); Study Completion 2023-06-23 (Estimated)

PRIMARY OUTCOMES:
Safety and effectivity - Incidence of study related adverse events | 24 weeks
  Incidence of study related adverse events which are defined as laboratory toxicities and clinical events that are possible, likely or definitely related to study treatment at any time from the infusion until week 24, including infusion related toxicity and any toxicity possibly related to CAR-BCMA T cells.
Engraftment | 2 years
  Duration of in vivo survival of CAR-BCMA T cells is defined as "engraftment". After 24 hours of infusion, the CAR-BCMA DNA sequence was detected by PCR according to the follow-up time point, until the result of any two consecutive tests was negative and recorded as the "engraftment endpoint" of CAR-BCMA T cells.

SECONDARY OUTCOMES:
Statistical parameter of efficacy assessment：PFS | 5 years
  Statistical parameter：Progression-free Survival (PFS)
Statistical parameter of efficacy assessment：DCR | 2 years
  Statistical parameter:Disease Control Rate (DCR)
Statistical parameter of efficacy assessment：ORR | 2 years
  Statistical parameter:Objective Remission Rate (ORR)
Statistical parameter of efficacy assessment：OS | 5 years
  Statistical parameter:Overall survival (OS)

OTHER OUTCOMES:
Number of DNA copies of CAR-BCMA T cells in tissue samples | 2 years
  Number of DNA copies of CAR-BCMA T cells in lymph node samples or bone marrow samples at regular intervals from 24 hours after the initial infusion.
Positive incidence of anti-drug antibody | 2 years
  Positive incidence of anti-BCMA anti-drug antibody (ADA).
Change of T cell subsets from baseline counts | 2 years
  Change of T cell subsets from baseline counts after infusion(Tcm, central memory T lymphocytes; Tem, effector memory T lymphocytes; Treg, regulatory T lymphocytes).

CONTACTS AND LOCATIONS:
Overall Officials: Jie Jin, MD, Principal Investigator — First Affiliated Hospital of Zhejiang University; Haitao Meng, MD, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No